CLINICAL TRIAL: NCT04730089
Title: Epidural Block Impairs Hypoxic Pulmonary Vasoconstriction During One-lung Ventilation: an Electrical Impedance Tomography- Based Prospective Observation Study
Brief Title: Epidural Block Impairs HPV During One-lung Ventilation: an EIT- Based Prospective Observation Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Ming Zhong, Professor, Shanghai Zhongshan Hospital
Other Study IDs: EB-EIT
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Epidural Block; Electrical Impedance Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Electrical impedance tomography — A bolus of 10ml 10% NaCl was injected during a respiratory pause (≥10s) through the central venous catheter.The results of arterial blood gas analysis and the data of EIT were collected before the first prone session (time baseline), the end of prone positioning (time P).

SUMMARY:
Define the effect of epidural block on HPV by EIT.

DETAILED DESCRIPTION:
Epidural block may affect the physiological mechanism of hypoxic pulmonary vasoconstriction, which is still poorly understood. Electrical impedance tomography might be helpful in establishing the hypoxemia etiology at bedside via combining regional ventilation and perfusion information.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years Existing central venous and arterial access Chest circumference 70 - 150 cm

Exclusion Criteria:

* Contraindication to central venous injection of 5 % sodium chloride (NaCl)

Contraindications of PulmoVista 500:

Patients with pacemakers, defibrillators or other electrically active implants Patients with damaged skin or impaired skin contact of the electrodes due to wound dressings Patients where the attachment of the patient belt could pose a risk to the patient, e.g. patients with spinal lesions or fractures Patients with uncontrolled body movements Extremely obese patients (BMI>50) Patients during pregnancy Patients with massive lung edema Use during electricity-based therapies, such as electrosurgery or electrocautery Use in the presence of strong magnetic fields Use in conjunction with other bioimpedance measurement devices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring thoracic surgery are given combined epidural anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Assess regional distribution of pulmonary perfusion | within 24 hours
  To evaluate the effect of epidural block on pulmonary blood flow distribution.
Assess oxygenation status | within 24 hours
  To evaluate the effect of epidural block by assessing regional distribution of pulmonary perfusion based on indicator dilution and changes at different points in time during varying states of regional ventilation will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhong, MD, phD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Y, Wei Y, Chen G, Wang Z, Fan Y, Wang J, Yang Y, Zhou D, Zhong M. The effects of thoracic epidural blockade on ventilation-perfusion matching during one-lung ventilation: An exploratory study. J Clin Anesth. 2024 Dec;99:111678. doi: 10.1016/j.jclinane.2024.111678. Epub 2024 Nov 6. PMID 39504921